CLINICAL TRIAL: NCT04897204
Title: A Prospective Randomized Controlled Study of Additonal Left Atrial Appendage Electrical Isolation in Catheter Ablation Combined With Left Atrial Appendage Occlusion of Persistent Atrial Fibrillation
Brief Title: Left Atrial Appendage Electrical Isolation in Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: ZHONGNANSHAN MEDICAL FOUNDATION OF GUANGDONG PROVINCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-21-004
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage; Left Atrial Appendage Occlusion; Catheter Ablation
Keywords: Left Atrial Appendage Electrical Isolation; Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Atrial Appendage Electrical Isolation with One-stop treatment of atrial fibrillation (Experimental): The patients received routine catheter ablation of atrial fibrillation with left atrial appendage occlusion and additional left atrial appendage electrical isolation operation.
  Interventions: Procedure: Additional left atrial appendage electrical isolation combined with catheter ablation and left atrial appendage occlusion
- One-stop treatment of atrial fibrillation (Other): The patients received routine catheter ablation of atrial fibrillation with left atrial appendage occlusion.
  Interventions: Procedure: Catheter ablation and left atrial appendage occlusion

INTERVENTIONS:
Procedure: Catheter ablation and left atrial appendage occlusion — The patients underwent routine pulmonary vein isolation and linear ablation and left atrial appendage occlusion.
  Arms: One-stop treatment of atrial fibrillation
Procedure: Additional left atrial appendage electrical isolation combined with catheter ablation and left atrial appendage occlusion — These patients underwent routine pulmonary vein isolation and linear ablation and left atrial appendage occlusion, combined with additional left atrial appendage occlusion.
  Arms: Left Atrial Appendage Electrical Isolation with One-stop treatment of atrial fibrillation

SUMMARY:
This project intends to enroll patients with persistent atrial fibrillation who are planning to undergo catheter ablation of atrial fibrillation. The two groups of patients were routinely performed atrial fibrillation pulmonary vein isolation and linear ablation with left atrial appendage occlusion. The experimental group received additional left atrial appendage electrical isolation before the left atrial appendage occlusion, and the control group did not perform left atrial appendage electrical isolation. We are intend to evaluate the safety and effectiveness of one-stop operation of left atrial appendage electrical isolation combined with left atrial appendage occlusion in the treatment of persistent atrial fibrillation.

DETAILED DESCRIPTION:
This project intends to enroll patients with persistent atrial fibrillation who are planned to undergo atrial fibrillation catheter ablation and left atrial appendage closure surgery, and randomly allocate them to the experimental group and the control group at a ratio of 1:1. The two groups of patients were routinely performed atrial fibrillation pulmonary vein isolation and linear ablation with left atrial appendage occlusion. The experimental group received additional left atrial appendage electrical isolation before the left atrial appendage occlusion, and the control group did not perform left atrial appendage electrical isolation. Follow-up for 1 year, compare the differences in the recurrence rate of atrial fibrillation between the two groups of patients, and further compare the differences in clinical events such as stroke, systemic embolism, hospitalization due to heart failure, and cardiovascular death.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old;
2. Symptomatic, non-valvular persistent atrial fibrillation (atrial fibrillation duration ≥ 1 week), and is ineffective to one or more anti-arrhythmic drugs;
3. CHA2DS2-VASc score ≥ 2 points;
4. The patient is ready to undergo atrial fibrillation catheter ablation and left atrial appendage closure surgery;
5. Provide an informed consent form that is willing to participate in the research, follow-up trials and evaluation procedures.

Exclusion Criteria:

1. Past left atrial appendage occlusion, atrial fibrillation catheter ablation or surgical ablation history;
2. There are plans for cardiac surgery within 90 days;
3. Stroke/transient ischemic attack occurred within 30 days;
4. Have had atrial septal defect repair or have an ASD/PFO occluder in the body;
5. Heart failure NYHA heart function grade IV;
6. LVEF<30%;
7. Combined with other serious diseases, the life expectancy is less than 2 years;
8. Within 6 months after cardiac revascularization or other cardiac surgery;
9. Women who are pregnant, breastfeeding, planning to become pregnant, or women of childbearing age who have not adopted reliable contraceptive methods;
10. Obviously abnormal liver and kidney function and coagulation function;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | one year after operation
  outside the 3-month blank period after surgery, ECG and Holter recorded rapid atrial arrhythmia greater than 30S.
Stroke/TIA | one year after operation
  Patients may have cerebral ischemia, such as sudden limb movement and sensory disturbance, aphasia, transient blindness in one eye, etc., disturbance of consciousness, or symptoms of vertebral artery ischemia, such as vertigo, tinnitus, hearing impairment, diplopia, Unsteady gait and difficulty swallowing, etc., patients may have obvious infarcts in the brain, which can be confirmed clinically by CT or MRI.
Systemic embolism | one year after operation
  The clinical manifestations or evidence of embolism in the blood vessels of the system, including renal artery, splenic artery, mesenteric artery, etc. during the follow-up of the patient, and relevant examinations can be used to confirm the diagnosis.
Hospitalization rate due to heart failure | one year after operation
  During the follow-up period, patients need hospitalization for heart failure, including acute heart failure, acute exacerbation of chronic heart failure, etc., which can be combined with clinical symptoms, signs, biochemical examinations (such as NT-proBNP) and cardiac ultrasound Wait for a clear diagnosis.
Cardiovascular death | one year after operation
  The death of a patient due to cardiac structure, function, coronary artery disease, and arrhythmia can be diagnosed in combination with clinical practice.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hylek EM, Go AS, Chang Y, Jensvold NG, Henault LE, Selby JV, Singer DE. Effect of intensity of oral anticoagulation on stroke severity and mortality in atrial fibrillation. N Engl J Med. 2003 Sep 11;349(11):1019-26. doi: 10.1056/NEJMoa022913. PMID 12968085
- [Result] Nyong J, Amit G, Adler AJ, Owolabi OO, Perel P, Prieto-Merino D, Lambiase P, Casas JP, Morillo CA. Efficacy and safety of ablation for people with non-paroxysmal atrial fibrillation. Cochrane Database Syst Rev. 2016 Nov 22;11(11):CD012088. doi: 10.1002/14651858.CD012088.pub2. PMID 27871122
- [Result] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Result] Di Biase L, Burkhardt JD, Mohanty P, Mohanty S, Sanchez JE, Trivedi C, Gunes M, Gokoglan Y, Gianni C, Horton RP, Themistoclakis S, Gallinghouse GJ, Bailey S, Zagrodzky JD, Hongo RH, Beheiry S, Santangeli P, Casella M, Dello Russo A, Al-Ahmad A, Hranitzky P, Lakkireddy D, Tondo C, Natale A. Left Atrial Appendage Isolation in Patients With Longstanding Persistent AF Undergoing Catheter Ablation: BELIEF Trial. J Am Coll Cardiol. 2016 Nov 1;68(18):1929-1940. doi: 10.1016/j.jacc.2016.07.770. PMID 27788847
- [Result] Romero J, Michaud GF, Avendano R, Briceno DF, Kumar S, Carlos Diaz J, Mohanty S, Trivedi C, Gianni C, Della Rocca D, Proietti R, Perrotta L, Bordignon S, Chun JKR, Schmidt B, Garcia M, Natale A, Di Biase L. Benefit of left atrial appendage electrical isolation for persistent and long-standing persistent atrial fibrillation: a systematic review and meta-analysis. Europace. 2018 Aug 1;20(8):1268-1278. doi: 10.1093/europace/eux372. PMID 29342299
- [Result] Fink T, Ouyang F, Heeger CH, Sciacca V, Reissmann B, Keelani A, Schutte C, Wohlmuth P, Maurer T, Rottner L, Eitel C, Eitel I, Rillig A, Metzner A, Kuck KH, Tilz RR, Vogler J. Management of thrombus formation after electrical isolation of the left atrial appendage in patients with atrial fibrillation. Europace. 2020 Sep 1;22(9):1358-1366. doi: 10.1093/europace/euaa174. PMID 32743641
- [Result] Kim YG, Shim J, Oh SK, Lee KN, Choi JI, Kim YH. Electrical isolation of the left atrial appendage increases the risk of ischemic stroke and transient ischemic attack regardless of postisolation flow velocity. Heart Rhythm. 2018 Dec;15(12):1746-1753. doi: 10.1016/j.hrthm.2018.09.012. PMID 30502771
- [Result] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Result] Belgaid DR, Khan Z, Zaidi M, Hobbs A. Prospective randomized evaluation of the watchman left atrial appendage closure device in patients with atrial fibrillation versus long-term warfarin therapy: The PREVAIL trial. Int J Cardiol. 2016 Sep 15;219:177-9. doi: 10.1016/j.ijcard.2016.06.041. Epub 2016 Jun 15. PMID 27343417
- [Result] Mo BF, Sun J, Zhang PP, Li W, Chen M, Yuan JL, Yu Y, Wang QS, Li YG. Combined Therapy of Catheter Ablation and Left Atrial Appendage Closure for Patients with Atrial Fibrillation: A Case-Control Study. J Interv Cardiol. 2020 Jun 25;2020:8615410. doi: 10.1155/2020/8615410. eCollection 2020. PMID 32669982
- [Result] Panikker S, Jarman JW, Virmani R, Kutys R, Haldar S, Lim E, Butcher C, Khan H, Mantziari L, Nicol E, Foran JP, Markides V, Wong T. Left Atrial Appendage Electrical Isolation and Concomitant Device Occlusion to Treat Persistent Atrial Fibrillation: A First-in-Human Safety, Feasibility, and Efficacy Study. Circ Arrhythm Electrophysiol. 2016 Jul;9(7):e003710. doi: 10.1161/CIRCEP.115.003710. PMID 27406602
- [Result] Yorgun H, Canpolat U, Kocyigit D, Coteli C, Evranos B, Aytemir K. Left atrial appendage isolation in addition to pulmonary vein isolation in persistent atrial fibrillation: one-year clinical outcome after cryoballoon-based ablation. Europace. 2017 May 1;19(5):758-768. doi: 10.1093/europace/eux005. PMID 28340073